CLINICAL TRIAL: NCT05038098
Title: Magnetic Sentinel Lymph Node Mapping in Gastric Cancer, Safety and Feasibility Clinical Trial
Brief Title: Magnetic Sentinel Lymph Node Mapping in Gastric Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0410; NCI-2021-08919 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0410 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-27; First posted 2021-09-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Gastric Adenocarcinoma
MeSH Terms: interventions — Gastrectomy; Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Cohort I (preoperative injection) (Experimental): Patients receive FerroTrace peritumorally within days 1-21. Patients then undergo gastrectomy and receive ICG peritumorally.
  Interventions: Procedure: Gastrectomy; Drug: Indocyanine Green; Other: Iron Conjugated Polymers in Saline Suspension
- Cohort II (intraoperative) (Experimental): Patients undergo gastrectomy and receive FerroTrace and ICG peritumorally during surgery.
  Interventions: Procedure: Gastrectomy; Drug: Indocyanine Green; Other: Iron Conjugated Polymers in Saline Suspension

INTERVENTIONS:
Procedure: Gastrectomy — Undergo surgery
  Other Names: Gastric Resection
Drug: Indocyanine Green — Given peritumorally
  Other Names: ICG
Other: Iron Conjugated Polymers in Saline Suspension — Given peritumorally
  Other Names: FerroTrace

SUMMARY:
This phase I finds out the possible benefits and/or side effects of using magnetic tracer FerroTrace and the fluorescent dye indocyanine green to identify the lymph nodes that cancer is most likely to have spread to in patients with gastric cancer that are undergoing gastrectomy. Using FerroTrace in combination with the indocyanine green dye may help researchers better detect the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess safety by assessing short term toxicity associated with the gastric injection of the novel magnetic tracer.

SECONDARY OBJECTIVES:

I. To determine the feasibility of sentinel lymph node (SLN) imaging and mapping using novel magnetic nanoparticles (iron conjugated polymers in saline suspension [FerroTrace]) for gastric cancer, and to determine whether pre-operative injection, intra-operative injection, or both are feasible.

II. To test the validity of this procedure by correlating sentinel lymph nodes (SLN) to predict pathologic Lymph node (LN)-positive status i.e., will a negative SLN accurately predict the negativity of the other LNs? III. To determine the diagnostic value of additional hematoxylin and eosin (H&E) sections and immunohistochemistry to assess sentinel lymph nodes compared to routine assessment with one H&E stain alone.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I (PREOPERATIVE INJECTION): Patients receive FerroTrace peritumorally within days 1-21. Patients then undergo gastrectomy and receive indocyanine green (ICG) peritumorally.

COHORT II (INTRAOPERATIVE INJECTION): Patients undergo gastrectomy and receive FerroTrace and ICG peritumorally during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing to provide informed consent
* Biopsy proven gastric cancer, undergoing curative-intent gastrectomy
* No distant metastases
* Pathologic diagnosis of gastric adenocarcinoma
* Pre-treatment endoscopic measurement of less than or equal to 4 cm in diameter of the gastric cancer

Exclusion Criteria:

* Contraindications to surgery +/- adjuvant therapy
* Allergy or intolerance to iron oxide compounds
* Allergy or intolerance to iodides
* Iron overload disorder
* Pregnant or lactating women*

  * Use of contraception is required for females during the study. Male patients who are sexually active with a female of childbearing potential are allowed for study enrollment and will not require use of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Safety of endoscopic peritumoral gastric injection of FerroTrace | Within 24 hours of the FerroTrace injection
  The Bayesian method by Thall et al. will be applied for interim toxicity monitoring. Toxicities are defined as any grade III or greater toxicities attributable to FerroTrace injection, which occur within 24 hours of the injection. Will summarize the rate of adverse events (AEs) in all patients and by cohort, along with the exact 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Naruhiko Ikoma, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org